CLINICAL TRIAL: NCT04316026
Title: Effectiveness of Shock Wave Therapy to Treat Upper Limb Spasticity in Hemiparetic Patients
Brief Title: Effectiveness of Shock Wave Therapy for Upper Limb Spasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/27MAR/151
Record Dates: First submitted 2020-01-07; First posted 2020-03-20 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): group receiving shock wave therapy
  Interventions: Device: shock wave therapy
- control group (Sham Comparator): sham shock wave therapy
  Interventions: Device: shock wave therapy

INTERVENTIONS:
Device: shock wave therapy — Shockwave therapy is a non-invasive treatment creating a series of low energy acoustic wave pulsations that are directly applied through the skin via a gel medium

SUMMARY:
Introduction: Shock wave therapy (SWT) has a potential interest to treat spasticity. However, the pathophysiology of this treatment remains unknown. Some authors assert that it is effective on spasticity itself, while others suggest that it acts more on fibrosis.

Method: this study will assess the effectiveness of radial SWT to treat wrist and finger flexors stiffness in stroke patients, comparing subacute spastic patients (< 12 months) with chronic patients presenting muscle contractures (> 12 months). Forty-eight stroke patients (24 in the subacute phase and 24 in the chronic phase) will be included. One real and one sham sessions of SWT will be performed with a 2-week interval. The order of the sessions will be randomized. Motor control, stiffness and spasticity will be assessed with clinical and objective measures, just after and just before each session, by a blind assessor. The targeted muscles will be flexor carpi radialis, flexor carpi ulnaris and flexor digitorum profundus, and will be the same for the two session.

ELIGIBILITY:
Inclusion Criteria:

* History of cerebral lesion
* Wrist spasticity ≥ 1+/4 on the Modified Ashworth Scale
* Wrist spasticity ≥ 2/4 on the Tardieu Scale
* Passive dorsal extension of the wrist ≥ 10°

Exclusion Criteria:

* Botulinum toxin injection in the upper limb in the past three months
* History of wrist arthrodesis
* Myopathy
* Treatment with oral anticoagulants or coagulation disease
* Tumor or infection of the paretic upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Before (baseline) and 5 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  Clinical assessment of spasticity for wrist and fingers flexors, score from 0 to 4 (a higher score representing a greater spasticity)
Tardieu scale | Before (baseline) and 5 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  Clinical assessment of spasticity for wrist and fingers flexors; score from 0 to 4 (a higher score representing a greater spasticity)

SECONDARY OUTCOMES:
objective measure of elastic and viscous stiffness of the wrist, expressed in N.m.rad | Before (baseline) and 5 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  electronic oscillatory device for stiffness measurement
objective measure of muscle stiffness | Before (baseline) and 10 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  Myoton measurement device
manual goniometer | Before (baseline) and 10 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  Passive measure of joint range of motion
Medical Research Council muscle testing | Before (baseline) and 25 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  strength assessment; score from 0 to 5 (a higher score representing a greater strength)
Isokinetic dynamometer | Before (baseline) and 15 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  objective measure of muscle stiffness at the wrist
H reflex | Before (baseline) and 5 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  electrophysiological assessment of the H reflex (motoneuronal excitability)
Box and block test | Before (baseline) and 30 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  measure of manual ability
Fugl Meyer Assessment - computerized adaptive testing | Before (baseline) and 25 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  neurological impairment
Abilhand scale | Before (baseline) and 45 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  PROMS on bimanual activities; a higher score represents a better manual ability
Wolff Motor Function Test | Before (baseline) and 35 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  manual activities
Visual Analog Scale | Before (baseline) and 45 minutes (post-treatment) after each of the two sessions (sham or real SWT)
  patient self-assessment of overall effectiveness of SWT; score from 0 to 4 (a higher score representing a greater improvement)

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan Stoquart, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No